CLINICAL TRIAL: NCT02958098
Title: My Research Legacy Pilot Study
Status: Terminated | Type: Observational
Why Stopped: Sponsor withdrew funding
Sponsor: American Heart Association (Other)
Responsible Party: Sponsor
Other Study IDs: My Research Legacy Pilot Study
Record Dates: First submitted 2016-11-04; First posted 2016-11-08 (Estimated); Last update posted 2021-03-08 (Actual); Status verified 2021-03

CONDITIONS: Myocardial Infarction; Stroke; Cardiomyopathy, Dilated; Systolic Heart Failure; Atrial Fibrillation; Aortic Dissection
Keywords: myocardial infarction; stroke; dilated cardiomyopathy; systolic heart failure; atrial fibrillation; aortic dissection; wearable devices; genomic sequencing
MeSH Terms: conditions — Myocardial Infarction; Stroke; Cardiomyopathy, Dilated; Heart Failure, Systolic; Atrial Fibrillation; Aortic Dissection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (5):
- Myocardial infarction: Individuals with myocardial infarction before age 50 years.
- Stroke: Individuals with stroke before age 50 years
- Aortic dissection: Individuals with aortic dissection before age 50 years
- Systolic heart failure: Individuals with systolic heart failure/dilated cardiomyopathy before age 50 years.
- Atrial fibrillation: Individuals with atrial fibrillation before age 50 years

SUMMARY:
The My Research Legacy Pilot Study will establish a participant registry that collects self-reported health data and answers to online survey questions about individual daily choices, diets, and exercise; data from wearable devices; and, (optional) data from genome sequencing analysis. Individuals under the age of 50 who meet eligibility criteria will answer questions using the American Heart Association's (AHA) Life's Simple 7™ My Life Check v4.0 three times over the course of 6 months and transmit data from a Fitbit Charge 2 device. All other individuals who are interested in the study and meet entry criteria may also enroll.

DETAILED DESCRIPTION:
2,000 Participant My Research Legacy Pilot Study

1. Day 0 - Enroll online, complete AHA's Life's Simple 7™ Survey Prospective participants will enroll in the research initiative via the My Research Legacy website (MyResearchLegacy.org). They will go through an online process in which they will answer brief, pre-qualifying questions before consenting to participate in the study.

   * Participants will attest to their age and US residence, and will provide a self-reported diagnosis of cardiovascular disease (myocardial infarction, atrial fibrillation, aortic dissection, systolic congestive heart failure/cardiomyopathy) and/or stroke.
   * Eligible participants will read and sign an online consent form.
   * Within the participant console, the participants will answer AHA's Life's Simple 7™ My Life Check v4.0 assessment.
   * Participants will be asked during the consent process if they will consent to provide medical records relevant to their diagnosis.
2. Day 90 Complete AHA's Life's Simple 7™ My Life Check v4.0 assessment; Start transmission from the Fitbit Charge 2.
3. Online Survey and contact Day 180 after enrollment, participants will receive an email requesting that they visit the participant console to repeat AHA's Life's Simple 7™ My Life Check v4.0 survey. Participants also have the option of determining whether or not they want to be contacted for future studies.

ELIGIBILITY:
Inclusion Criteria:

1. Age > or = to 18 years but < 50 years.
2. History of one (or more) of the following:

   1. Myocardial infarction
   2. Stroke
   3. Aortic dissection
   4. Systolic heart failure/cardiomyopathy
   5. Atrial fibrillation
3. Individuals of any age > or = 18 years who don't have above medical conditions but want to participate in the study.
4. Access to a computer and/or cell phone with internet access.

Exclusion Criteria:

1. Unwillingness to sign informed consent
2. No access to a computer and/or cell phone with internet access.

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All individuals equal to or older than 18 years but younger than 50 years of age who have a history of, or have, an aortic dissection; or systolic heart failure/cardiomyopathy; or atrial fibrillation; or myocardial infarction; or stroke. All other individuals equal to or older than 18 years who don't meet the above health criteria but are interested in the study.
Sampling Method: Non-Probability Sample
Enrollment: 2267 (Actual)
Dates: Start 2016-11-11 (Actual); Primary Completion 2018-10-30 (Actual); Study Completion 2018-10-30 (Actual)

PRIMARY OUTCOMES:
study retention | 6 months
  continues to engage with study after 6 months

SECONDARY OUTCOMES:
Change in answers to AHA's Life's Simple 7™ My Life Check v4.0 | 6 months
  answers to second and other surveys
Duration of time Fitbit Charge 2 used by participants | 6 months
  recorded time
Change in Fitbit Charge 2 step count | 6 months
  recorded steps
Percent of individuals that initiate but don't complete online process | 6 months
  number that start but don't finish first surveys
Activity duration | 6 months
  Daily, weekly, monthly activity from Fitbit Charge 2

CONTACTS AND LOCATIONS:
Overall Officials: Jane A Leopold, MD, Principal Investigator — American Heart Association

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be made available to other researchers.

REFERENCES:
- [Derived] Leopold JA, Antman EM. Digital health device measured sleep duration and ideal cardiovascular health: an observational study. BMC Cardiovasc Disord. 2021 Oct 14;21(1):497. doi: 10.1186/s12872-021-02284-z. PMID 34649522